CLINICAL TRIAL: NCT04744688
Title: Changes in Coagulation in Colorectal Cancer Patients Undergoing Surgical Treatment
Acronym: CONTEST
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-212-20
Record Dates: First submitted 2021-01-04; First posted 2021-02-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2020-12

CONDITIONS: Peritoneal Metastases; Peritoneal Carcinomatosis; Colorectal Neoplasms Malignant; Intestinal Neoplasms; Cytoreductive Surgery; Venous Thromboembolism; Bleeding; Laparoscopic Surgery; Coagulation; Surgical Procedures, Operative; Postoperative Complications; Laparoscopy; Minimally Invasive Surgical Procedures; Surgical Oncology
Keywords: Bleeding; Venous thromboembolism; Coagulation; Cancer surgery; Thromboprophylaxis; Colorectal cancer; Cancer; Peritoneal metastases; Postoperative complications; Rectal cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Colonic Neoplasms; Intestinal Neoplasms; Venous Thromboembolism; Hemorrhage; Thrombosis; Postoperative Complications; Colorectal Neoplasms; Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 48 cytoreductive surgery with HIPEC patients: 48 patients with peritoneal metastases from colorectal cancer undergoing cytoreductive surgery with HIPEC (cytoreductive surgery with HIPEC patients)
- 48 minimally invasive patients: 48 rectal cancer patients undergoing minimally invasive rectal cancer resection

SUMMARY:
Cytoreductive surgery with hyperthermic intraperitoneal chemotherapy (HIPEC) has prolonged the survival substantially for selected patients with peritoneal metastases from colorectal cancer.Bleeding and thromboembolic disease have been reported as postoperative complications related to this advanced open surgical treatment. However, perioperative changes in coagulation and fibrinolysis are only sparsely reported in the literature.The mainstay of treatment with curative intend of none-advanced colorectal cancer is minimally invasive laparoscopic surgery followed by adjuvant chemotherapy. The approach is considered associated with a lower risk of thromboembolic disease than open surgery. Despite differences in extent of surgery and thromboembolic risk the same extended thromboprophylaxis regimen for 28 days is currently prescribed to patients undergoing cytoreductive surgery with HIPEC as well as minimally invasive rectal cancer resection. This study aims to investigate all parts of the coagulation system and fibrinolysis, and thereby thromboembolic risk and potential bleeding in two groups of patients with different extent of surgical trauma: 1) Colorectal cancer patients undergoing cytoreductive surgery with HIPEC and 2) rectal cancer patients undergoing minimal invasive rectal cancer resection. Our hypothesis is that patients undergoing cytoreductive surgery with HIPEC are exposed to more aggravated alterations of coagulation and fibrinolysis than patients undergoing minimally invasive rectal cancer resection.

ELIGIBILITY:
Inclusion Criteria:

Cytoreductive surgery with HIPEC patients:

* Able to give informed consent
* Age ≥ 18 years
* Diagnosed with peritoneal metastases from colorectal cancer
* Planned to undergo cytoreductive surgery with HIPEC

Minimally invasive rectal cancer patients:

* Able to give informed consent
* Age ≥ 18 years
* Diagnosed with rectal cancer
* Planned to undergo minimal invasive rectal cancer resection with one of: total mesorectal excision, partial mesorectal excision or abdominoperineal excision

Exclusion Criteria (both groups):

* Thromboembolic event within 90 days before surgery
* Secondary malignancy within previous 5 years or concomitant, except non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include patients with peritoneal metastases from colorectal cancer undergoing cytoreductive surgery with HIPEC and rectal cancer patients undergoing minimally invasive rectal cancer resection. Patients will be identified at the outpatient clinic and undergo surgical treatment at the Department of Surgery, Aarhus University Hospital, Denmark.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
The difference between changes in concentration of prothrombin fragment 1+2. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.

SECONDARY OUTCOMES:
The difference between changes in platelet concentration from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of immature platelets from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of plasma selectin from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in activated partial thromboplastin time "APTT" (seconds) from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in international normalized ratio "INR" (seconds) from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of plasma fibrinogen from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of coagulation factor VIII from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of von wildebrand factor from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of thrombin-antithrombin complex from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in thrombin generation before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
  Thrombin generation will be measured by:
  Lagtime (min), time to peak (min), peak thrombin (nM) and endogenous thrombin potential (nM*min).
The difference between changes of fibrin clot structure from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference between changes of fibrin clot structure from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
  Fibrin clot structure will be measured by clot maximum, absorbance (arbitrary units), network density, lysis time (seconds), lysis area (balance between clot formation and lysis).
The difference between changes in concentration of plasminogen activator inhibitor-1 from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of fibrin d-dimer from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in global hemostasis by Rotational thromboelastometry (ROTEM) from before surgery to the end of surgery (both groups) | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery (both groups).
  ROTEM will include EXTEM, INTEM, FIBTEM, and APTEM by clotting time (seconds), clot formation time (seconds), alpha-angle (degrees), amplitude 10 min after clotting time (mm), maximum clot firmness (mm), lysis index 30 min after clotting time (mm), maximum lysis (mm).
The difference between changes in concentration of syndecan-1 from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of sE-selectin from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of soluble thrombomodulin. from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of hemoglobin from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration of leucocytes from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection.
The difference between changes in concentration C-reactive protein (CRP) from before surgery to the end of surgery in cytoreductive surgery with HIPEC patients and patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from before surgery to the end of surgery in cytoreductive surgery.
The difference between changes in concentration of prothrombin fragment 1+2. from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end HIPEC.
The difference between changes in platelet concentration from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of immature platelets from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in activated partial thromboplastin time "aPTT" (seconds) from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in activated international normalized ratio "INR" (seconds) from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of plasma fibrinogen from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of coagulation factor VIII from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of von wildebrand factor from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of thrombin-antithrombin complex from the end of cytoreductive surgery to the end HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in thrombin generation from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC. Thrombin generation will be measured by: Lagtime (min), time to peak (min), peak thrombin (nM) and endogenous thrombin potential (nM*min).
The difference between changes of fibrin clot structure from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC. Fibrin clot structure will be measured by clot maximum, absorbance (arbitrary units), network density, lysis time (seconds), lysis area (balance between clot formation and lysis).
The difference between changes in concentration of plasminogen activator inhibitor-1 from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of fibrin d-dimer from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of global hemostasis measured by Rotational thromboelastometry (ROTEM) from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery to the end HIPEC.
  ROTEM will include EXTEM, INTEM, FIBTEM, and APTEM by clotting time (seconds), clot formation time (seconds), alpha-angle (degrees), amplitude 10 min after clotting time (mm), maximum clot firmness (mm), lysis index 30 min after clotting time (mm), maximum lysis (mm).
The difference between changes in concentration of syndecan-1 from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end HIPEC.
The difference between changes in concentration of sE-selectin from the end of cytoreductive surgery to the end of HIPEC | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of soluble thrombomodulin from the end of cytoreductive surgery to the end of HIPEC | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of hemoglobin from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of leucocytes from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years.
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
The difference between changes in concentration of C-reactive protein (CRP) from the end of cytoreductive surgery to the end of HIPEC. | Data will be analyzed, assessed, and presented within three years
  The difference will be measured in blood samples from the end of cytoreductive surgery (before HIPEC) to the end of HIPEC.
Incidence of deep vein thrombosis measured by doppler ultrasonography in colorectal cancer patients undergoing minimally invasive rectal cancer resection. | Data will be analyzed, assessed, and presented within three years
  Bilateral doppler ultrasonography of the veins in the lower extremities.The scan will be performed within the postoperative period from day 3 to day 7.
Incidence of deep venous thrombosis measured by doppler ultrasonography in colorectal cancer patients undergoing cytoreductive surgery with HIPEC | Data will be analyzed, assessed, and presented within three years
  Bilateral doppler ultrasonography of the veins in the lower extremities.The scan will be performed within the postoperative period from day 3 to day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, MD, PhD, Principal Investigator — Thrombosis and Haemostasis Research Unit, Department of Clinical Biochemistry, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Thrombosis and Haemostasis Research Unit, Department for Clinical Biochemistry, Aarhus University Hospital, Aarhus N